CLINICAL TRIAL: NCT06751589
Title: Pilot Weight Loss Intervention With Dual GIP/GLP-1 Receptor Agonist Therapy in Patients With Endometrial Cancer and Obesity, Overweight, With or Without Diabetes
Brief Title: A Study of a Weight Loss Intervention in People With Endometrial Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-331
Record Dates: First submitted 2024-12-20; First posted 2024-12-30 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Endometrial Cancer
Keywords: tirzepatide; semaglutide; dual GIP/GLP-1 receptor; obesity; overweight; diabetes; stage I-III endometrial cancer
MeSH Terms: conditions — Endometrial Neoplasms; Obesity; Overweight; Diabetes Mellitus | interventions — Tirzepatide

STUDY DESIGN:
Intervention Model Description: This is a single institution, single arm pilot study among Endometrial Cancer (EC) patients with obesity/overweight or diabetes undergoing chemotherapy to determine the feasibility and and preliminary efficacy of a weight loss intervention with weekly SC tirzepatide.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- tirzepatide (Experimental): Patients will meet with the study endocrinologist during screening and be prescribed SC tirzepatide 2.5 mg administered using a pre-filled injector once weekly for 4 weeks and then increase to 5 mg once weekly. If insurance does not cover tirzepatide, the GLP-1 agonist semaglutide (Wegovy, Ozempic) initiated at 0.25 mg weekly SC may be substituted if deemed appropriate by the study PI.
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — 2.5 mg administered using a pre-filled injector once weekly for 4 weeks and then increase to 5 mg once weekly.

SUMMARY:
The researchers are doing this study is to find out whether tirzepatide and semaglutide are practical (feasible) for weight management and blood sugar control for endometrial cancer patients undergoing chemotherapy. The researchers will also look at participants' experience with the study drug, the safety of taking the study drug while receiving chemotherapy, and changes in weight, body fat composition, and blood pressure of participants.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* Obesity (defined as BMI ≥ 30 kg/m2) OR Overweight (defined as BMI ≥ 27 kg/m2) with presence of ≥1 weight related comorbid condition OR a diagnosis of Type 2 Diabetes Mellitus with BMI ≥ 25 kg/m2
* Type 2 Diabetes Mellitus is defined as known history of Type 2 diabetes, HbA1c ≥ 6.5%, fasting blood glucose ≥126 mg/dL on 2 occasions, or random blood glucose ≥ 200 mg/dL with signs and symptoms of diabetes mellitus (weight loss, fatigue, polyuria, polydipsia, vision changes)
* Patients with new diagnosis of stage I-III endometrial cancer
* Completed surgery with TH/BSO with no gross residual disease
* Recommended to undergo curative intent adjuvant chemotherapy at MSK with carboplatin and paclitaxel with or without intravaginal radiation OR cisplatin and concurrent radiation followed by carboplatin and paclitaxel. Patients may consent prior to and up to 3 weeks after the first cycle of chemotherapy.
* Patients with the following histologic epithelial cell types are eligible: endometrioid adenocarcinoma, serous adenocarcinoma, carcinosarcoma, undifferentiated carcinoma/de-differentiated, clear cell adenocarcinoma, mixed epithelial carcinoma, adenocarcinoma not otherwise specified (N.O.S.), and mucinous adenocarcinoma.
* Patient has adequate organ function, as defined by the following laboratory values:

  1. Creatinine clearance (per Cockcroft-Gault formula) ≥30 mL/min
  2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3.0 × ULN.
  3. Total serum bilirubin ≤ 1.5 × ULN except for patients with Gilbert's syndrome who may be included if the total serum bilirubin is ≤3.0 × ULN or direct bilirubin ≤ 1.5 × ULN.
* Insurance approval for tirzepatide or semaglutide (alternative) or willingness to pay out-of-pocket for tirzepatide or semaglutide (alternative) for duration of study period
* Patients must be capable and willing to learn how to self-inject study drug, as required for this protocol (visually impaired persons who are not able to perform the injections must have the assistance of a sighted individual trained to inject study drug; persons with physical limitations who are not able to perform the injections must have the assistance of an individual trained to inject study drug) and administer study drug injection (or receive an injection from a trained individual if visually impaired or with physical limitations)
* Not pregnant and not nursing
* English speaking or a family member or caregiver who speaks English and is able to assist with smart phone or tablet based Keenoa app or paper dietary recall handout (if no access to smart phone or tablet).

Exclusion Criteria:

* Known Type 1 diabetes
* Known GAD, Islet Cell, or Zn Transporter 8 antibodies
* History of gastroparesis
* High risk for aspiration
* Active or history of chronic or acute pancreatitis
* History of elevated calcitonin
* Personal or family history of Medullary Thyroid Carcinoma with Multiple Endocrine Neoplasia-2 syndrome
* Patients with a prior surgical, endoscopic, and/or device-based therapy (for example, mucosal ablation, gastric artery embolization, intragastric balloon and duodenojejunal bypass sleeve) for obesity within the past two years
* Patients with removal of device-based therapy for obesity within the last 6 months
* Current GIP/GLP-1 or GLP-1 receptor agonist use or prior intolerance of GIP/GLP-1 or GLP-1 receptor agonist
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Known intolerance to study drug(s) or any of the excipients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Endometrial cancer
Enrollment: 36 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
percentage of patients that complete treatment | 1 year
  measured by the percentage of patients that complete at least 70% of weekly doses, specifically 17 out of 24 weekly doses.

SECONDARY OUTCOMES:
frequency of gastrointestinal adverse events | up to 24 2weeks
  as graded by CTCAE 5.0 that are attributable to the study treatment (tirzepatide) and occur during the on-treatment period from baseline initiation of the intervention to the end of study

CONTACTS AND LOCATIONS:
Overall Officials: Angela Green, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm